CLINICAL TRIAL: NCT00571168
Title: Randomised, Placebo Controlled, Single-center, Double-blind Clinical Trial to Investigate Efficacy and Safety of Aprepitant Combined With Kevatril and Dexamethasone Versus Placebo Combined With Kevatril and Dexamethasone in Prevention of Acute and Delayed High-dose Chemotherapy-induced Nausea and Vomiting in Subjects With Multiple Myeloma Receiving an Autologous Peripheral Blood Stemcell Transplantation.
Brief Title: Efficacy and Safety of Aprepitant in Subjects With Multiple Myeloma During and After High-dose Chemotherapy
Acronym: EmNa
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Gerlinde Egerer / MD, University of Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EmNa (2001-004956-38); EudraCT-No: 2004-004956-38
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Multiple Myeloma
Keywords: chemotherapy induced nausea and vomiting; autologous peripheral blood stemcell transplantation; high dose chemotherapy
MeSH Terms: conditions — Multiple Myeloma; Vomiting | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Aprepitant plus standard therapy (Kevatril + Dexamethason) on day 1-4
  Interventions: Drug: Emend
- B (Placebo Comparator): Placebo plus standard therapy (Kevatril + Dexamethason) on day 1-4
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Emend — 125 mg/d on day 1; 80 mg/d on day 2-4
  Arms: A
Drug: Placebo — Placebo capsules on day 1-4
  Arms: B

SUMMARY:
1. Scientific background In patients with multiple myeloma high-dose chemotherapy followed by autologous stemcell transplantation is preferred to conventional therapy, since the superiority in respect to complete remission, complete remission duration, event-free survival and overall survival has been proven within well controlled clinical trials (Fassas et al., 2002; Goldschmidt et al., 2003).

   Nausea and vomiting are well known and the most distressing side-effects of a high dose chemotherapy regimen. The administration of selective 5-HT3-receptor antagonists (5-HT3 RAs) in combination with a corticosteroid (= antiemetic standard therapy) is effective for the prevention of those adverse effects in 70 to 80 % of patients. However, 25 to 40 % of the patients still suffer from vomiting and nausea in the delayed phase of the chemotherapy. Superior protection could be achieved with the addition of Aprepitant (EMEND®) to the antiemetic standard therapy in acute and delayed phases of highly emetogenic chemotherapies. The enhanced antiemetic protection can be maintained over multiple chemotherapy-cycles to an extent superior to that of standard therapy alone (de Wit et al., 2003).

   Furthermore addition of Aprepitant (EMEND®) to standard therapy was generally well tolerated and the impact of chemotherapy-induced nausea and vomiting (CINV) on daily life was significantly reduced (Hesketh et al., 2003; Dando & Perry, 2004).
2. Trial Rationale Aprepitant (EMEND®) is a selective high-affinity receptor antagonist of human substance P/neurokinin-1 (NK1) and has been shown to inhibit emesis induced by cytotoxic chemotherapeutic agents and augments the antiemetic activity of 5-HT3 RAs (e.g. Granisetron, Ondansetron) and corticosteroids (e.g. Dexamethasone). Thus Aprepitant (EMEND®) in addition to antiemetic standard therapy has been shown to possess powerful superior protection and has been reported in several clinical trials to significantly improve both acute and delayed CINV.

The aim of this study is to evaluate, during and up to 7 days after high-dose chemotherapy with Melphalan (moderate emetogenic drug) followed by autologous peripheral blood stemcell transplantation, an antiemetic treatment regimen in respect to efficacy and safety in patients with multiple myeloma. To the best of our knowledge effects of Aprepitant on Melphalan induced CINV have never been investigated.

ELIGIBILITY:
Inclusion Criteria:

* Men and women >/= 18 years
* Patients with multiple myeloma receiving high-dose chemotherapy (Melphalan) and autologous peripheral stemcell transplantation
* Signed informed consent

Exclusion Criteria:

* Patients suffering from nausea and vomiting during the last 12 hours prior to planned high-dose chemotherapy
* Patients receiving antiemetics 24 hours prior to planned high-dose chemotherapy
* Intake of steroids
* History of hypersensitivity to the investigational product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational product
* Simultaneous intake of pimozide, terfenadine, astemizole
* Pregnant or nursing woman
* Mental condition rendering the subject incapable to understand the nature, scope and possible consequences of the trial
* Expected non-compliance in completing the subject´s diary and FLIE-score

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Estimated)
Dates: Start 2005-07; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Overall complete response (no emesis and no rescue therapy) | During and post chemotherapy (0-120 h)

SECONDARY OUTCOMES:
Complete response acute/delayed phase | During and post chemotherapy (0-120h)
Vomiting event rate | During and post chemotherapy (0-120h)
No emesis (FLIE-Score) | During and post chemotherapy (0-120h)
No (significant) nausea (VAS < 5 mm;(< 25 mm)) | During and post chemotherapy (0-120h)
No rescue therapy | During and post chemotherapy (0-120h)
Total control (no emesis, no nausea, no rescue therapy) | During and post chemotherapy (0-120h)
No impact on daily life | During and post chemotherapy (0-120h)
AEs | During and post chemotherapy (0-120h)

CONTACTS AND LOCATIONS:
Overall Officials: Gerlinde Egerer, MD, Principal Investigator — University Hospital of Heidelberg; Im Neuenheimer Feld 410; 69120 Heidelberg/ Germany
Locations (1):
- University Hospital of Heidelberg, Department V, Heidelberg, Germany

REFERENCES:
- [Derived] Schmitt T, Goldschmidt H, Neben K, Freiberger A, Husing J, Gronkowski M, Thalheimer M, Pelzl le H, Mikus G, Burhenne J, Ho AD, Egerer G. Aprepitant, granisetron, and dexamethasone for prevention of chemotherapy-induced nausea and vomiting after high-dose melphalan in autologous transplantation for multiple myeloma: results of a randomized, placebo-controlled phase III trial. J Clin Oncol. 2014 Oct 20;32(30):3413-20. doi: 10.1200/JCO.2013.55.0095. Epub 2014 Sep 15. PMID 25225424